CLINICAL TRIAL: NCT00903357
Title: A Double Blind, Randomized, Crossover Study to Compare the Effectiveness of Montelukast on Atopic Dermatitis in Koreans
Brief Title: The Effectiveness of Montelukast on Atopic Dermatitis in Koreans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pyun BokYang (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Pyun BokYang, Professor, Soonchunhyang University Hospital
Organization: Soonchunhyang University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: schallergy
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Results first posted 2012-09-13 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Montelukast
MeSH Terms: conditions — Dermatitis, Atopic | interventions — montelukast; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Montelukast first, then placebo (Experimental): The group received active medication (montelukast 4 mg or 5mg once daily) for 8 weeks followed by a crossover to 8 weeks of placebo after 2-weeks washout period.
  Interventions: Drug: Montelukast first, then placebo; Drug: Placebo first, then Montelukast
- Placebo first, then Montelukast (Experimental): The group received placebo medication (ascorbic acid) for 8 weeks followed by a crossover to 8 weeks of active medication (montelukast 4 mg or 5mg once daily) after 2-weeks washout period.
  Interventions: Drug: Montelukast first, then placebo; Drug: Placebo first, then Montelukast

INTERVENTIONS:
Drug: Montelukast first, then placebo — Patients in "Montelukast first, then placebo" will receive 4 mg of montelukast under the age of 6 years (5 mg of montelukast at 6 years) once daily for 8 weeks. And after 2 weeks wash-out period, they will receive chewable ascorbic acid placebo for 8 weeks. Patients in "Placebo first, then Montelukast" are received chewable ascorbic acid placebo for 8 weeks. And after 2 weeks wash-out period, they will receive 4 mg of montelukast under the age of 6 years (5 mg of montelukast at 6 years) once daily for 8 weeks.
  Other Names: SINGULAIR
Drug: Placebo first, then Montelukast — Patients in "Montelukast first, then placebo" will receive 4 mg of montelukast under the age of 6 years (5 mg of montelukast at 6 years) once daily for 8 weeks. And after 2 weeks wash-out period, they will receive chewable ascorbic acid placebo for 8 weeks. Patients in "Placebo first, then Montelukast" are received chewable ascorbic acid placebo for 8 weeks. And after 2 weeks wash-out period, they will receive 4 mg of montelukast under the age of 6 years (5 mg of montelukast at 6 years) once daily for 8 weeks.
  Other Names: Ascorbic acid

SUMMARY:
The purpose of this study is to assess the clinical effectiveness of Montelukast in children (2~6 years old) with atopic dermatitis and identify the pathophysiologic background of Montelukast on the role of modulating the atopic dermatitis measured by urinary Leukotriene 4 (LTE4) and Eosinophil protein X(EDN).

DETAILED DESCRIPTION:
Leukotriene B4 (LTB4) and the cysteinyl-leukotrienes LTC4, LTD4 and LTE4 are potent proinflammatory mediators derived from arachidonic acid through the 5- lipoxygenase pathway. They are secreted from eosinophils and other inflammatory cells such as mast cells and macrophages. The primary action of leukotrienes includes contraction of human airway muscle, chemotaxis, and increased vascular permeability, with secondary effects of inhibiting allergen-induced early and late responses. Several in vivo and in vitro studies suggest a role for cysteinyl leukotrienes in the pathogenesis of atopic dermatitis and there is a rationale for the use of pharmacological agents to antagonize their effects in the treatment of atopic dermatitis. Levels of LTE4 measured in urine (Urinary-LTE4) may be a useful measure of whole-body cysteinyl-leukotriene production in vivo, because that LTE4 is a stable urinary metabolite of LTC4 and LTD4. Urinary-LTE4 has been measured in individuals with atopic dermatitis, but in small-scale studies, and the results are conflicting.

ELIGIBILITY:
Inclusion Criteria:

* The ages of 2 to 6 years old, 54 children with moderate to severe atopic dermatitis diagnosed by the criteria of Haniffin and Rajka were included in the study.
* Volunteer children with moderate to severe atopic dermatitis were recruited from the Pediatric Allergy and respiratory Center of the SoonChunHyang University Hospital (Seoul, Korea). At the time of recruitment, written consent was obtained. The ethical committee at the SoonChunHyang University Hospital approved the trial.
* Volunteers who agreed by their parents.
* The severity of their disease was assessed by modified SCORAD index.

Exclusion Criteria:

* Too severe atopic dermatitis defined as the sum of scores is 80 and above by SCORAD index.
* A history of liver disease; allergy to montelukast or cross-reacting medication; use of phenobarbital, phenytoin or rifampicin.
* Patients on systemic steroids, immune-suppression or Korean herbal medicine during the previous 6 weeks.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bok Yang Pyun, M.D., PhD., Study Chair — Pediatric Allergy & Respiratory Center, Department of Pediatrics, Soonchunhyang University Hospital
Locations (1):
- Pediatric Allergy & Respiratory Center, Department of Pediatrics, Soonchunhyang University Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Childrens(2~6 years old) with moderate to severe atopic dermatitis recruited from the Pediatric Allergy and respiratory Center of the SoonChunHyang University Hospital (Seoul, Korea).
Pre-assignment Details: 54 participants recruited.
Groups:
- Montelukast First, Then Placebo: Montelukast(4mg or 5mg) once daily in first intervention period and placebo(chewable ascorbic acid) once daily in second intervention period (after washout period).
- Placebo First, Then Montelukast: Placebo(chewable ascorbic acid) once daily in first intervention period and Montelukast(4mg or 5mg) once daily in second intervention period (after washout period).
Period: First Intervention
Arm/Group | Montelukast First, Then Placebo | Placebo First, Then Montelukast
Started | 27 | 27
Completed | 22 | 23
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Flu | 0 | 1
Period: Wash Out Period of 2 Weeks
Arm/Group | Montelukast First, Then Placebo | Placebo First, Then Montelukast
Started | 22 | 23
Completed | 22 | 22
Not Completed | 0 | 1
Not completed — Flu | 0 | 1
Period: Second Intervention
Arm/Group | Montelukast First, Then Placebo | Placebo First, Then Montelukast
Started | 22 | 22
Completed | 21 | 22
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive Montelukast first and placebo first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: months] | 46.0 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 27
Severity of atopic dermatitis [Number; unit: participants] — Severity of atopic dermatitis using SCORAD index. Moderate : 15~40, Severe : >40.
  participants
    moderate | 26
    severe | 28

OUTCOME MEASURES:

1. Primary Outcome: Changes in SCORAD Index
Description: Changes of SCORAD(SCORing Atopic Dermatitis) index after taking Montelukast or placebo drug. SCORAD calculation: Extent(%)/5 + 7*Intensity/2 + subjective symptoms (minimum score 0, maximum score 103) (SCORAD index >40: severe, 15-40:moderate, <15: mild)
Time Frame: 18 weeks after patient recruitment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Montelukast Sodium: Changes of SCORAD index after taking Montelukast Sodium. Patients were randomized to receive either montelukast(4 mg for under the age of 6 years, 5mg for 6 years and over) once daily or a chewable ascorbic acid placebo, which was comparable in size and color to the study drug for 8 weeks and cross-over for 8 weeks after 2 weeks wash-out period. We have collected data of SCORAD index before and after taking Montelukst Sodium in both group(Montelukast first, then placebo, and Placebo first, then Montelukast)
- Placebo Drug: Changes of SCORAD index after taking Placebo drug. Patients were randomized to receive either montelukast(4 mg for under the age of 6 years, 5mg for 6 years and over) once daily or a chewable ascorbic acid placebo, which was comparable in size and color to the study drug for 8 weeks and cross-over for 8 weeks after 2 weeks wash-out period. We have collected data of SCORAD index before and after taking placebo drug in both group(Montelukast first, then placebo, and Placebo first, then Montelukast)
Arm/Group | Montelukast Sodium | Placebo Drug
Number analyzed (Participants) | 43 | 43
units on a scale | -3.0 (11.2) | -5.7 (11.3)

2. Primary Outcome: Changes in Urinary LTE4
Description: Changes of Urinary LTE4(Leukotrien E4) after taking Montelukast or placebo drug. Urinary LTE4 levels were measured using an enzyme-linked immunoassay (ELISA) (Cayman Chemical, Michigan, USA) and the intra-assay and inter-assay variations were 7.4 ± 2.1 and 12.4 ± 7.8, respectively. Minimum value : 0 Maximum vlaue: 1000 pg/ml.
Time Frame: 18 weeks after patient recruitment
Measure: Mean (Standard Deviation); unit: Urinary LTE4 (pg/ml)
Groups:
- Montelukast Sodium: Changes of Urine LTE4 after taking Montelukast Sodium. Patients were randomized to receive either montelukast(4 mg for under the age of 6 years, 5mg for 6 years and over) once daily or a chewable ascorbic acid placebo, which was comparable in size and color to the study drug for 8 weeks and cross-over for 8 weeks after 2 weeks wash-out period. We have collected data of urinary LTE4 before and after taking Montelukst Sodium in both group(Montelukast first, then placebo, and Placebo first, then Montelukast)
- Placebo Drug: Changes of Urine LTE4 after taking Placebo drug. Patients were randomized to receive either montelukast(4 mg for under the age of 6 years, 5mg for 6 years and over) once daily or a chewable ascorbic acid placebo, which was comparable in size and color to the study drug for 8 weeks and cross-over for 8 weeks after 2 weeks wash-out period. We have collected data of urinary LTE4 before and after taking placebo drug in both group(Montelukast first, then placebo, and Placebo first, then Montelukast)
Arm/Group | Montelukast Sodium | Placebo Drug
Number analyzed (Participants) | 43 | 43
Urinary LTE4 (pg/ml) | -65.9 (556.2) | 87.7 (618.3)

3. Primary Outcome: Changes in Urinary EDN
Description: Changes of Urinary EDN(Eosinophil Derived Neurotoxin) after taking Montelukast or placebo drug. Urinary EDN levels were measured using an ELISA (MBL, Woburn, MA, USA) and the intra-assay and inter-assay variations were 3.0 ± 0.5 and 7.7 ± 1.5, respectively. Minimum value: 0, Maximum value: 2040 ng/ml.
Time Frame: 18 weeks after participants recruitment
Measure: Mean (Standard Deviation); unit: Urine EDN (ng/ml)
Groups:
- Montelukast Sodium: Changes of Urine EDN after taking Montelukast Sodium. Patients were randomized to receive either montelukast(4 mg for under the age of 6 years, 5mg for 6 years and over) once daily or a chewable ascorbic acid placebo, which was comparable in size and color to the study drug for 8 weeks and cross-over for 8 weeks after 2 weeks wash-out period. We have collected data of urinary EDN before and after taking Montelukast sodium in both group(Montelukast first, then placebo, and Placebo first, then Montelukast)
- Placebo Drug: Changes of Urine EDN after taking Placebo drug. Patients were randomized to receive either montelukast(4 mg for under the age of 6 years, 5mg for 6 years and over) once daily or a chewable ascorbic acid placebo, which was comparable in size and color to the study drug for 8 weeks and cross-over for 8 weeks after 2 weeks wash-out period. We have collected data of urinary EDN before and after taking placebo drug in both group(Montelukast first, then placebo, and Placebo first, then Montelukast)
Arm/Group | Montelukast Sodium | Placebo Drug
Number analyzed (Participants) | 43 | 43
Urine EDN (ng/ml) | 37.0 (1008.6) | -195.8 (916.7)

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- Montelukast Sodium: Montelukast sodium(4mg or 5mg) administered once daily in either first intervention period or second intervention period.
- Placebo Drug: Placebo drug administered once daily in either first intervention period or second intervention period.
Arm/Group | Montelukast Sodium | Placebo Drug
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less